CLINICAL TRIAL: NCT02784340
Title: Comparison of Local and Intra Venous Dexamethasone on Post Operative Pain and Recovery After Caeseream Section
Brief Title: Local and Intravenous Dexamethasone on Post Operative Pain a After CS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, Assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 148
Record Dates: First submitted 2016-05-20; First posted 2016-05-27 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Postoperative Pain
Keywords: Postoperative pain; dexamethasone; cesarean section
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexamethasone; dexamethasone 21-phosphate; Sodium Chloride; Fluid Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- IV dexamethasone (Active Comparator): 40 women received 16 mg Dexamethasone IV drip.
  Interventions: Drug: Dexamethasone; Drug: Bupivicaine and Fentany; Device: 25G spinal needles
- Local dexamethasone (Active Comparator): 40 women received 16 mg Dexamethasone subcutaneous injection around the caesarean section scar after skin closure
  Interventions: Drug: Dexamethasone; Drug: Bupivicaine and Fentany; Device: 25G spinal needles
- placebo (Placebo Comparator): Placebo in the form of IV fluids 500 cc saline infusion
  Interventions: Drug: Saline (IV fluids); Drug: Bupivicaine and Fentany; Device: 25G spinal needles

INTERVENTIONS:
Drug: Dexamethasone — 16 mg Dexamethasone IV drip
  Other Names: dexamethasone sodium phosphate. EIPICO pharmaceutical, Egypt
  Arms: IV dexamethasone
Drug: Dexamethasone — 16 mg Dexamethasone subcutaneous injection around the caesarean section scar after skin closure
  Other Names: dexamethasone sodium phosphate USP 8mg/2ml amp. EIPICO pharmaceutical, Egypt
  Arms: Local dexamethasone
Drug: Saline (IV fluids) — IV fluids 500 cc saline infusion
  Other Names: saline infusion
  Arms: placebo
Drug: Bupivicaine and Fentany
Device: 25G spinal needles

SUMMARY:
A Prospective, randomized study conducted on 120 pregnant women attending the labour wards in Kasr Al Ainy and Fayoum maternity hospitals from May 2014 to December 2015. All participants were scheduled for elective cesarean section under spinal anaesthesia and were randomly divided into 3 equal groups. Group 1(40 women) received 16 mg Dexamethasone IV drip. Group II (40 women) received 16 mg Dexamethasone subcutaneous injection around the caesarean section scar after skin closure and Group III received Placebo in the form of IV fluids 500 cc saline infusion. All cases were followed up for 48 hours for assessment of level of pain by using a 10-cm visual analog scale (VAS). Primary outcome parameters were VAS score and the need for additional analgesics. Other parameters were hemodynamic changes and occurrence of side effects or complications

DETAILED DESCRIPTION:
The patients were subjected to history taking, including age, parity, menstrual history for verification of gestational age and medical history for confirmation of inclusion and exclusion criteria. Full general and abdominal and obstetric examinations were done. Investigations including complete blood picture, liver functions and coagulation profile to exclude those not fitting with the above listed criteria. Ultrasound was done to assess gestational age.

Patients were checked for coagulation abnormalities. Large gauge (18G) cannula was inserted in cephalic or ante cubital veins. Patients were preloaded with HAES- steril 6% (hydroxyl ethyl starch) Fresenius. Or, preloaded with ringer's lactate 20 ml/kg. Patients were positioned in the sitting position for spinal anaesthesia and sterilization of the back was done using Betadine. L3-L4 space was determined for the insertion of spinal needle. Then 25G spinal needle was used to perform a single shot spinal anaesthesia using 10mg of 0.5% hyperbaric Bupivicaine and Fentanyl 20 micrograms.

All surgeons had close surgical skills and used the same technique transverse lower segment incision.

The procedure is then completed using traction on cord to deliver the placenta, exteriorization of uterus, closure of uterine incision in 2 layers, closure of both visceral and parietal peritoneum, closure of rectus sheath, no subcutaneous closure and finally subcuticular skin closure. Follow up for all cases for 48 hours. Primary outcome parameters were VAS score and the need for additional analgesics. Other parameters were hemodynamic changes and occurrence of side effects or complications.

ELIGIBILITY:
Inclusion Criteria:

* All participants were scheduled for elective cesarean section under spinal anaesthesia

Exclusion Criteria:

* Women with neurological disorders
* Psychologically disturbed
* Those with uncontrolled hypertension, Diabetes Mellitus, peptic ulcer, liver cirrhosis or glaucoma
* Women with systemic infections
* Allergy to Dexamethasone
* Contraindications to spinal anaesthesia

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2014-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
VAS score visual acoustic score | 48 hours after CS
  Subjective description of the pain using questionaire

SECONDARY OUTCOMES:
need for additional analgesics | 48 hours after CS
Blood pressure | 48 hours after CS

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Kasr Alainy medical school

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maged AM, Deeb WS, Elbaradie S, Elzayat AR, Metwally AA, Hamed M, Shaker A. Comparison of local and intra venous dexamethasone on post operative pain and recovery after caeseream section. A randomized controlled trial. Taiwan J Obstet Gynecol. 2018 Jun;57(3):346-350. doi: 10.1016/j.tjog.2018.04.004. PMID 29880162